CLINICAL TRIAL: NCT05364346
Title: The HAPPY Study: Holistic Approach to Pregnancy and the First Postpartum Year
Brief Title: HAPPY Study: Holistic Approach to Pregnancy and the First Postpartum Year
Acronym: HAPPY
Status: Completed | Type: Observational
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, prof.dr. Victor J Pop, Prof.dr. Victor JM Pop, Tilburg University
Other Study IDs: HAPPY2014
Record Dates: First submitted 2014-02-13; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Pregnancy
Keywords: pregnancy-related symptoms; psychological distress; thyroid function; postpartum well-being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood analysis of thyroid function and HCG. TSH, FT4, TPO-Ab, and HCG will be measured in Li-heparin plasma using electrochemoluminescence assays.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women in the area of South-East Brabant, The Netherlands

SUMMARY:
The HAPPY study is a large prospective longitudinal cohort study in which pregnant women (N≈2,500) are followed during the entire pregnancy and the whole first year postpartum. The study collects a substantial amount of psychological and biological data investigating all kinds of determinants that might interfere with general well-being during pregnancy and postpartum, with special attention to the effect of maternal mood, pregnancy-related somatic symptoms (including nausea and vomiting (NVP) and carpal tunnel syndrome (CTS) symptoms), thyroid function, and human chorionic gonadotropin (HCG) on pregnancy outcome of mother and foetus.

The primary aim of HAPPY concerning pregnancy is to measure the prevalence and changes of biological signs and symptoms over time, with special focus on NVP and CTS. Both a psychological and a biological model will be tested to explain the variance of (severe) NVP and CTS symptoms.

Also, the occurrence of maternal distress (anxiety and depression) will be assessed during different trimesters. Secondly, we will measure the changes in thyroid functioning over time during pregnancy and investigate a possible independent effect of thyroid dysfunction on foetal development as assessed by a standardized ultrasound protocol at 18-22 weeks gestation. Moreover, a possible independent effect of thyroid dysfunction on maternal mood will be investigated as well as on obstetric outcome including abnormal foetal position at term, the prevalence of preterm birth (< 37 weeks of gestation) and its possible causes such as preterm premature rupture of membranes (PPROM), the occurrence of pre-eclampsia and other obstetric complications.

With regard to the postpartum period, the primary aim is to investigate the effect of chronic depression during pregnancy on postpartum recovery. Secondary outcome is the impact of thyroid autoimmune disease on postpartum depression. Tertiary outcome is the relation between psychological determinants and initiating and continuation of breastfeeding.

DETAILED DESCRIPTION:
Recruitment: Dutch-speaking Caucasian women (or third generation women of other ethnic groups) who have their first prenatal visit are eligible to participate in the study from the early beginning of their pregnancy. Eligible pregnant women (and their partner) receive written and oral information about the study at their first prenatal visit. If women decide to participate, written informed consent will be obtained. Written informed consent includes participation in the study and inclusion of all obstetric data from the medical record form of the community midwife and obstetrician (including ultrasound data), a detailed delivery description and neonatal condition, and data of newborn screening (heel prick test).

Sample size calculation: The total amount of pregnancies in the area of the 17 community midwife practices is about 5,000 per year. With 10-15% non-Caucasian, 10-15% early abortion rate and 1.7% gemelli pregnancies, approximately 3,700 pregnant women will be eligible annually. Based on previous pregnancy-related research experiences of the last 20 years in this area, the response rate is expected to be high (70%) especially when no additional blood tests or interventions have to be performed. This will result in about 2,600 inclusions annually. During pregnancy, the rate of women moving outside the area is in general low which means that a number of 2,500 women are expected to finish the study protocol until delivery. After a pilot period of three months followed by a running-in period of three months, it is estimated that all midwife practices will collaborate within six months. Therefore, the period of recruitment will take 18 months to include 2,600 women.

Because different types of events with different prevalence rates might interfere with the sample size needed for appropriate statistics, the number of 2,500 women is estimated to meet the standard epidemiological criteria. With 2,500 participants, the following numbers of abnormal events are estimated to be found: 108 women with a foetus in breech position (4.3%), 185 preterm births (7.4%), 450 women (18%) will develop depression during pregnancy and 325-475 women (13-19%) will develop postpartum depression during the first postpartum year. According to thyroid function, the investigators will find 200 (8%) women with elevated titres of thyroid peroxidase antibodies (TPO-Ab) and 100 with thyrotrophin (TSH) levels > 2.5 IU/l. These numbers will allow statistical analysis with sufficient power. With an expected prevalence rate of 4-10% (breech, preterm birth, TPO antibodies, TSH > 2.5), a significance level of 5% and a power of 80%, 1,500-2,140 women need to be included (depending on the expected prevalence rate). In order to anticipate on (low) drop out, 2,600 women will be included.

Data collection:

* Questionnaires (eight questionnaires during the period between 12 weeks gestation and 12 months postpartum)
* Obstetric record form
* Standardized 20 weeks ultrasound (SEO)
* Blood analysis of thyroid function and HCG. The Primary Care laboratory of Eindhoven (Diagnostics voor U) will be responsible for collection of the blood samples and the ultrasounds. The Laboratory of clinical chemistry and haematology of the Máxima Medical Centre Veldhoven is responsible for analysis of TSH, free-thyroxin (FT4), TPO-Ab and HCG and storage of the blood samples. Since the additional tube of blood will be drawn during the regular blood assessment (which already needs a venipuncture), and the umbilical cord and the placenta normally are thrown away for destruction after birth, it can be stated that there are no additional interventions performed to either mother or the newborn within the HAPPY study.

Ethical approval: The HAPPY study is approved by the Ethical Board of Tilburg University (with special attention to the type of questionnaires that are used) and has been evaluated by the Medical Ethical Committee of the Máxima Medical Centre Veldhoven. Because all additional blood samples were obtained during regular blood assessments as part of regular obstetric care, the board confirmed that no additional approval of a medical committee was needed.

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 18 years
* Caucasian women (or third generation women of other ethnic groups) who are able to complete Dutch questionnaires
* Singleton pregnancy
* Term of gestation at inclusion < 14 weeks only if the women did not have had their standard blood assessment

Exclusion Criteria:

* Gemelli pregnancy
* Endocrine disorder
* Use of thyroid medication
* Severe psychiatric disease (schizophrenia, borderline, or bipolar disorder)
* HIV
* Drug or alcohol addiction problems
* Any other disease resulting in treatment with drugs that are potentially adverse for the foetus and need careful follow-up during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 2269 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy-related signs and symptoms during pregnancy | 12, 22, 32 weeks of gestation and 1 week postpartum
  * Prevalences and changes of pregnancy-related symptoms like nausea and vomiting (NVP) and carpal tunnel syndrome (CTS) during pregnancy
  * Relation between psychological determinants and NVP
  * Relation between thyroid function, HCG and NVP
  * Relation between thyroid function and CTS
Maternal distress | 12, 22, 32 weeks of gestation and postpartum at 1 week, 6 weeks, 4 months, 8 months and 1 year
  * Prevalences and changes in maternal distress (anxiety and depression) during pregnancy and the first year postpartum
  * Relation between psychological determinants and initiating and continuation of breastfeeding

SECONDARY OUTCOMES:
Thyroid function | 10-12 weeks an 26-30 weeks of gestation
  * changes in thyroid functioning over time during pregnancy
  * investigate a possible independent effect of thyroid dysfunction on foetal development as assessed by a standardized ultrasound protocol at 18-22 weeks gestation
  * effect of thyroid dysfunction on maternal mood
  * effect of thyroid dysfunction on obstetric outcome
  * impact of thyroid autoimmune disease on postpartum depression

CONTACTS AND LOCATIONS:
Overall Officials: Victor J Pop, MD, PhD, Principal Investigator — Tilburg University